CLINICAL TRIAL: NCT04559178
Title: Impact of Intraoperative Fluid Challenges Administration on Macro and Microcirculation in Patients Undergoing High-risk Abdominal Surgery and Situated in the Gray Zone of Pulse Pressure Variation
Brief Title: Fluid Challenges and Microcirculation
Acronym: FC
Status: Terminated | Type: Observational
Why Stopped: too difficult to measure sublingual microcirculation continuously during a fluid challenge
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Study Director, Erasme University Hospital
Other Study IDs: P2020/338 / B4062020000092
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Fluid challenge — fluid challenge administration when patient is in the gray zone

SUMMARY:
The goal of this prospective observational study is to assess the impact of fluid challenge administration on macro and microcirculation in patients situated in the gray zone during a high risk abdominal surgery

DETAILED DESCRIPTION:
Fluid optimization is a key goal in anesthesia. It allows to titrate fluid bolus based on flow variables or dynamic parameters of fluid responsiveness (pulse pressure variation (PPV) or stroke volume variation (SVV)).

When PPV or SVV is above 13%, the patient will usually respond to a bolus of fluid while when PPV or SVV is below 9%, the patient will normally not respond to it. Between 9% and 13%, it is a gray zone where the effect of a fluid bolus is uncertain.

The overall goal of fluid bolus administration is of course to optimize macrocirculation (stroke volume and cardiac output) but also (and probably more importantly) end organ tissue perfusion. However, regional tissue perfusion is not widely monitored during surgery. However, we do have some monitoring tools to assess microcirculation at the bedside.

Investigation of microcirculation in addition to macro circulation may allow clinicians to know if a patient situated in the gray zone may or not increase microcirculation variables while macrocirculation variables are well known to be of little value to predict fluid responsiveness.

The goal of this study is to assess microcirculation variables in patients situated in the gray zone (PPV between 9%-13%), and to assess macro and microcirculation responses to a standardized fluid challenge of 4 ml/kg of a balanced crystalloid solution.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a high-risk abdominal surgery
* Patients equipped with a minimally invasive cardiac output monitoring device in order to optimize fluid administration

Exclusion Criteria:

* Atrial fibrillation
* Ejection fraction <40%

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for a high-risk abdominal surgery and equipped with a minimally uncalibrated pulse contour analysis monitoring device as part of their anesthetic care.
  All patients will have the hemodynamic monintoring to assess macrocirculation and sublingual microcirculation.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Microvascular flow index | day 0
  Comparison of this index before and after the fluid challenge

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre JOOSTEN, MD PhD, Study Director — ERASME; Alexandra Colesnicenco, MD, Principal Investigator — ERASME
Locations (1):
- Bicetre hospital, Le Kremlin-Bicêtre, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided